CLINICAL TRIAL: NCT01579877
Title: Efficacy of Yukmijihwang-tang on Xerostomia in the Elderly: A Randomized,Double-blind, Placebo-controlled, Two-center Trial
Brief Title: Treatment of Xerostomia by Herbal Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jin-sung Kim, Full professor, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KOMCIRB2011-28/KHNMC-OH-IRB20
Record Dates: First submitted 2012-04-13; First posted 2012-04-18 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Xerostomia
Keywords: Xerostomia; Yukmijihwang-tang; Yin-Deficiency; Visual analogue scale; Dry mouth symptom questionnaire
MeSH Terms: conditions — Xerostomia; Yin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yukmijihwang-tang (Experimental): Yukmijihwang-tang: Real herbal extract granule
  Interventions: Dietary Supplement: Herbal extract granule
- Yukmijihwang-tang_Placebo (Placebo Comparator): Yukmijihwang-tang_Placebo: Placebo herbal extract granule
  Interventions: Dietary Supplement: Placebo herbal extract granule

INTERVENTIONS:
Dietary Supplement: Herbal extract granule — The herbal extract granule, Yukmijihwang-tang granule, consists of 6 herbs. Ingredients: Rehmanniae Radix, Deoscoreae Radix, Corni Fructus, Hoelen, Alismatis Radix, Paeoniae Radicis Cortex. Dosage and frequency: 1 pack (3g), 3 packs per day (2 hours after morning, afternoon and evening meal)
  Other Names: Hexalong Granule
  Arms: Yukmijihwang-tang
Dietary Supplement: Placebo herbal extract granule — The Yukmijihwang-tang_Placebo has the same form, color and flavor as experimental intervention (Yukmijihwang-tang). The dosage, frequency and duration is also the same as experimental intervention (Yukmijihwang-tang).
  Other Names: Hexalong Granule Placebo
  Arms: Yukmijihwang-tang_Placebo

SUMMARY:
The aims of this study are to investigate the effect of famous herbal formula extract on xerostomia, and to determine whether this formula affect various xerostomia-related questionnaires, salivary flow rate, residual saliva and salivary tests.

DETAILED DESCRIPTION:
Xerostomia is a condition related to both decrease in the amount of saliva produced and a change in its composition, therefore causing dry mouth.It can cause severe decline in quality of life and up to date, there have been few effective treatments for xerostomia.

The purpose of the current trial is to investigate the effect of herbal extract granule named Yukmijihwang-tang (YMT) on dry mouth. The trial is a randomized, double-blinded, placebo-controlled, 2-arm, 2-centered study. Ninety-six patients with xerostomia will be randomly assigned to one of the 2 groups consisting of YMT or placebo. The assigned treatments will last for 8 weeks and the follow-up period will be 2 weeks.

The primary outcomes are Visual analogue scale (VAS) for xerostomia.

The present study is designed to examine the safety and efficacy of YMT on xerostomia. Our study provides the clinical evidence of a new therapeutic strategy for xerostomia.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 60 - 80
2. The visual analog scale for xerostomia must represent more than 4 points during 2wks prior to enrollment
3. One who has less than 0.3 ml/min of unstimulated salivary flow rate
4. One who has complained of xerostomia for at least 3months
5. One who is able to read, write, hear, see something
6. One who agree on not taking other therapies during experimental period
7. One who agree on consent form

Exclusion Criteria:

1. One who is taking the treatment for autoimmune disease such as sjogren's disease, rheumatic disease, systemic lupus erythematosus etc
2. One who has the history of taking radiotherapy on head and neck or history of organ transplantation
3. One who has severe mental illness such as depression
4. One who takes oriental medicine or health functional food within 2 wks before enrollment
5. One who takes the remedies on the purpose of relieving xerostomia such as pilocarpine, cevimeline, gargle solution, frequent gum use, intra oral devices and toothpaste etc.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for xerostomia | Visit 1(0week), Visit 2(4week), Visit 3(8week), Visit 4(10week)
  A 100 mm measurement instrument will be given to the patient and he will be instructed to indicate his severity of xerostomia in relation to the 2 extremes (0: no fatigue, 100: very severe fatigue).

SECONDARY OUTCOMES:
Unstimulated Salivary Flow Rate (USFR) and Stimulated salivary flow rate (SSFR) | Visit 1(0week), Visit 2(4week), Visit 3(8week), Visit 4(10week)
Residual saliva | Visit 1(0week), Visit 2(4week), Visit 3(8week), Visit 4(10week)
Salivary IgA, Chromogranin A, Cortisol | Visit 1(0week), Visit 3(8week)
Dry Mouth Symptom Questionnaire(DMSQ) | Visit 1(0week), Visit 2(4week), Visit 3(8week), Visit 4(10week)
  DMSQ is composed of 10 questions associated with the severity of xerostomia and various behaviors related to xerostomia

CONTACTS AND LOCATIONS:
Overall Officials: Jinsung Kim, doctorate, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Oriental Medicine Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Han G, Park JW, Ko SJ, Son J, Seon J, Kim J, Kim S, Yeo I, Ryu B, Kim J. Yukmijihwang-tang for the treatment of xerostomia in the elderly: study protocol for a randomized, double-blind, placebo-controlled, two-center trial. Trials. 2013 Sep 3;14:281. doi: 10.1186/1745-6215-14-281. PMID 24004451